CLINICAL TRIAL: NCT05310383
Title: Combination of Immune Checkpoint Inhibitors Tislelizumab and Radiotherapy for Recurrent, Metastatic and Persistent Advanced Cervical Cancer: A Single-arm, Single-center, Phase 2 Clinical Study
Brief Title: Tislelizumab and Radiotherapy for Recurrent Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMURADIO2
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Recurrent Cervical Carcinoma; Metastatic Cervical Carcinoma; Persistent Cervical Carcinoma; Radiotherapy; Immunotherapy; Anti-programmed Cell Death Receptor 1; Immune Checkpoint Inhibitors; Tislelizumab; Objective Response Rate; Survival Outcomes
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent cervical cancer (Experimental): Patients with recurrent, metastatic and persistent advanced cervical cancer
  Interventions: Combination Product: Tislelizumab plus radiotherapy

INTERVENTIONS:
Combination Product: Tislelizumab plus radiotherapy — During the period of radiotherapy, patients receiveTislelizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W). Tislelizumab 200mg q3W was administered for up to 35 cycles (up to approximately 2 years) after radiotherapy until disease progression or toxicity.

SUMMARY:
This study is a prospective, multicenter, phase II clinical trial to evaluate the efficacy and safety of albumin-bound paclitaxel plus bevacizumab for platinum-resistant recurrent epithelial ovarian cancer. Patients with platinum-resistant recurrent ovarian cancer who meet the inclusion criteria, and don't meet any of the exclusion criteria, are enrolled in the study. They will receive albumin-bound paclitaxel (260 mg/m2) and bevacizumab (7.5mg/kg) intravenously every 21 days. The total treatment periods are no more than 6 cycles. Treatment continue until disease progression, intolerable toxicity, or patient refusal. Objective response rates primary objective. Progression-free survival, overall survival, and safety are secondary objectives. The study will enroll a total of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates and signs informed consent
2. Aged 18 years of age or older
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 within 7 days prior to the first dose of study treatment
4. Has recurrent cervical cancer and controllable local treatment, indicating an indication for radiation therapy
5. Willing to accept concurrent radiotherapy combined with Tislelizumab
6. Has measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the local investigator
7. Has adequate organ function
8. Has expected survival time ≥3 months

Exclusion Criteria:

1. Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
2. Has a known history of Human Immunodeficiency Virus (HIV) infection，active Hepatitis virus infection and active tuberculosis (TB; Bacillus tuberculosis)
3. Has known active central nervous system (CNS) metastases and/or uncontrolled, untreated carcinomatous meningitis with elevated intracranial pressure
4. Has received a major surgery within 4 weeks prior to signing informed consent
5. Not suitable for radiotherapy
6. Reassessment of liver and kidney function and blood routine indexes after radiotherapy did not meet the above criteria
7. Did not meet the other requirements for inclusion by the investigator
8. Judged unqualified of the enrollment requirements by the researcher according to other conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-03-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  PFS defined as the time the duration from date of enrollment to the first documented disease progression, or death due to any cause, whichever occurs first.
Overall survival | 24 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause
Adverse Events | 24 months
  Adverse event (AE), Treatment emergent adverse event (TEAE), Serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China